CLINICAL TRIAL: NCT01139463
Title: Blood Lactate Levels in Patients Treated With Typical or Atypical Antipsychotics
Brief Title: Study of Blood Lactate Levels in Patients Treated With Antipsychotics
Status: Completed | Type: Observational
Sponsor: University of Split (Other)
Responsible Party: Trpimir Glavina, University of Split
Other Study IDs: 500-03/06-01/74, 2181-147-06
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Movement Disorders; Lactic Acidosis
Keywords: antipsychotics; lactates; side effects
MeSH Terms: conditions — Movement Disorders; Acidosis, Lactic | interventions — Haloperidol; Olanzapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Antipsychotic treatment: Patients were not taking any medications - apart from the prescribed antipsychotic - for a period of 1 month prior to the study with psychotic relapse or newly diagnosed psychotic disorder were recruited from psychiatric inpatient and outpatient clinics of the Split Clinical Hospital.
  Interventions: Drug: Haloperidol or olanzapine

INTERVENTIONS:
Drug: Haloperidol or olanzapine — Haloperidol tablet - 5 mg twice daily (morning and evening) by mouth Olanzapine tablet - 5 mg twice daily (morning and evening) by mouth
  Other Names: Haldol; Olzapin

SUMMARY:
Blood lactate levels in patients receiving typical or atypical antipsychotics have not been described in the literature.

The goal of this study is to assess the dynamics of lactate levels in the blood from typical or atypical antipsychotics not confounded by prior antipsychotic treatments, the investigators conducted a prospective study of lactate levels in patients receiving antipsychotic medication. The investigators hypothesized that 6 months of treatment with haloperidol or olanzapine would result in a change in blood lactate levels and extrapyramidal side effects.

DETAILED DESCRIPTION:
The aim of this study was to compare the blood lactate levels in patients receiving typical or atypical antipsychotics.

Subjects included sixty patients with psychotic disorder were assigned to treatment for 6 months with haloperidol (typical antipsychotic), N=30 or olanzapine (atypical antipsychotic), N=30. Blood lactate levels, other metabolic parameters, and scores on the extrapyramidal symptom rating scale (ESRS) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 - 50 years
* Not taking any antipsychotic medication 1 month prior to the study
* Diagnosed psychotic disorder

Exclusion Criteria:

* Female
* Tobacco use
* Diabetes mellitus
* Baseline lactate blood level over 2.0 mmol/L

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population consists of patients from the psychiatric inpatient and outpatient sections of a primary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Blood lactate levels | 1 month
Blood lactate levels | 3 months
Blood lactate levels | 6 months

SECONDARY OUTCOMES:
Extrapyramidal side effects | 1 month
  The extrapyramidal symptom rating scale (ESRS) was used for assessment of four types of antipsychotic induced movement disorders: parkinsonism, akathisia, dystonia, and tardive dyskinesia referred to as extrapyramidal side effects in this study.
Extrapyramidal side effects | 3 months
  The extrapyramidal symptom rating scale (ESRS) was used for assessment of four types of antipsychotic induced movement disorders: parkinsonism, akathisia, dystonia, and tardive dyskinesia referred to as extrapyramidal side effects in this study.
Extrapyramidal side effects | 6 months
  The extrapyramidal symptom rating scale (ESRS) was used for assessment of four types of antipsychotic induced movement disorders: parkinsonism, akathisia, dystonia, and tardive dyskinesia referred to as extrapyramidal side effects in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Trpimir Glavina, MD, Principal Investigator — University of Split
Locations (1):
- Split Clinical Hospital Center, Split, Croatia

REFERENCES:
- [Derived] Glavina T, Mrass D, Dodig T, Glavina G, Pranic S, Uglesic B. Blood lactate levels in patients receiving first- or second- generation antipsychotics. Croat Med J. 2011 Feb;52(1):41-7. doi: 10.3325/cmj.2011.52.41. PMID 21328719